CLINICAL TRIAL: NCT04116645
Title: Time Frame for GBS Screening
Status: Withdrawn | Type: Observational
Why Stopped: This study would not add any new information
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dana Vitner MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0251-19-RMB
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: GBS; Group B Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: singleton pregnancies
  Interventions: Other: genital and rectal swab
- Group 2: Twin pregnancies
  Interventions: Other: genital and rectal swab

INTERVENTIONS:
Other: genital and rectal swab — 6. Swabs for GBS culture should be obtained, ideally before digital examination or use of lubricants, from both the lower vagina (vaginal introitus) and rectum (insert swab through the anal sphincter) to achieve maximum sensitivity. Either two swabs (one for each site) or a single swab can be used; one swab is more cost saving. The swabs will be obtained by the patient herself after appropriate instruction or by the provider healthcare, as studies have shown equivalent sensitivity between the healthcare provider and the patient herself.

SUMMARY:
All pregnant women prenatally being followed up or admitted at Rambam HealthCare Campus, Haifa, Israel are potential participants in the study. If a patient is agreeable, the nurse/physician/research coordinator will obtain informed consent.

Once informed consent is obtained, the patient can be swabbed for GBS. The swabs will be obtained at the routine follow-up at the clinic at 30, 32 and 35 weeks' gestation.

If a patient is found to have a positive GBS culture at 35 weeks, she will receive antibiotic treatment during labour according to the protocol.

GBS swabs taken at delivery will be compared to previous swabs taken at an earlier gestational age in order to evaluate sensitivity, specificity, positive and negative predictive values of GBS swabs at each week of gestation and to determine the value of our primary hypothesis.

DETAILED DESCRIPTION:
1. All pregnant women prenatally being followed up or admitted at Rambam HealthCare Campus, Haifa, Israel are potential participants in the study.
2. Most high-risk pregnant women have their routine follow ups every two weeks or less from the beginning of the third trimester (between 28 and 32 weeks' gestation).
3. The nurse/physician/research coordinator in the clinic will discuss the trial with those women. If a patient is agreeable, the nurse/physician/research coordinator will obtain informed consent.
4. Once informed consent is obtained, the patient can be swabbed for GBS.
5. The swabs will be obtained at the routine follow-up at the clinic at 30, 32 and 35 weeks' gestation. Then, they will be handed to the nurse/physician/research coordinator and transferred to the lab for analysis.
6. Swabs for GBS culture should be obtained, ideally before digital examination or use of lubricants, from both the lower vagina (vaginal introitus) and rectum (insert swab through the anal sphincter) to achieve maximum sensitivity. Either two swabs (one for each site) or a single swab can be used; one swab is more cost saving. The swabs will be obtained by the patient herself after appropriate instruction as studies have shown equivalent sensitivity between the healthcare provider and the patient herself20.
7. The swabs should be placed promptly into non-nutrient transport media (eg, Amies or Stuart's without charcoal) and transported at room temperature (in temperate climates) or refrigerated. The swabs are then transferred to a selective enrichment broth at a laboratory experienced in the isolation of GBS, incubated overnight at 37ºC, and subcultured onto blood agar plates. Cultures require 24 to 48 hours to show positive results. It takes 48 hours to definitively exclude GBS20.
8. The swabs will be kept for seven days, then will be removed by environmental services for their discard process.
9. A log of all patients who meet all inclusion criteria and agreed to participate in the trial will be maintained, recording the date and gestational age. GBS swab results will also be recorded. We will only reveal the results from the 35 weeks' screening to the main care provider of the patient as part of the common practice. We will not provide the other screening results, neither to the patient nor to their physician.
10. If a patient is found to have a positive GBS culture at 35 weeks, she will receive antibiotic treatment during labour according to the protocol.
11. GBS swabs taken at delivery will be compared to previous swabs taken at an earlier gestational age in order to evaluate sensitivity, specificity, positive and negative predictive values of GBS swabs at each week of gestation and to determine the value of our primary hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women that are being followed up prenatally or admitted at Rambam HealthCare Campus, Haifa, Israel and are planning to deliver there.
2. Women at gestational age 300/7 or less.

Exclusion Criteria:

1. Age 18 and under.
2. Women with previous delivery of an infant affected by GBS disease.
3. Women with known bacteriuria in the current pregnancy.
4. Women whom are planning not to deliver at Rambam HealthCare Campus.
5. Women who will not consent to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to conduct an open label prospective trial of all women with a singleton pregnancy which will be screened for GBS in four different time-points during their pregnancy, from 30 weeks' gestation up to delivery - 30, 32, 35 weeks' gestational age and at delivery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Determination of the best timing for GBS screening. | 10 weeks for each woman from the first swab to the last (at delivery)
  When is the best time to swab for GBS and what is the percentage of women with the same swab results at 30 or 32 weeks' gestation and at delivery

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive values of GBS swabs in each week of gestation | 10 weeks fpr each woman

CONTACTS AND LOCATIONS:
Overall Officials: Dana Vitner, M.D, Principal Investigator — vitnerdana@gmail.com

IPD SHARING:
Plan to Share IPD: No